CLINICAL TRIAL: NCT02159404
Title: Seasonal Differences in Nasal Mucus Proteome and Impact of Immunotherapy
Brief Title: Nasal Mucus Proteome and Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Tomazic Peter Valentin, MD, Medical Doctor, Medical University of Graz
Other Study IDs: ProtOmicsSeasons01; KLI 425-B23 (Other Grant/Funding Number: Austrian Science Fund (FWF))
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Allergic Rhinoconjunctivitis
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Allergic Rhinoconjunctivitis: Patients with diagnosed Allergic Rhinoconjunctivitis
  Interventions: Biological: Immunotherapy
- Healthy controls

INTERVENTIONS:
Biological: Immunotherapy
  Groups: Allergic Rhinoconjunctivitis

SUMMARY:
Nasal mucus as first line defense barrier of the nasal mucosa contains a variety of proteins that act as functional units. We recently showed that the nasal mucus proteome between allergic rhinitis patients and healthy controls is significantly altered.

The aim of the present project is to show changes in nasal mucus proteome between allergic rhinitis patients and healthy controls over the pollen and non pollen season and to further determine whether and if so how the proteome changes under immunotherapy. Patients and healthy controls will be enrolled at two time points namely during the pollen season and out of the pollen season. Statistical differences will be determined within the groups and between the groups as well as impact of immunotherapy on patients undergoing therapy.

Mucus will be collected with a special suction device equipped with a mucus trap. Then, proteomic analysis will be performed by LC MS/MS mass spectrometry. Database search will identify distinct proteins and their function, origin etc. will be annotated. Protein groups will be analyzed through pathway enrichment and cluster analysis. Furthermore, mechanisms of immunotherapy in responders and success or failure of therapy could be determined. These could lead to the identification of potential biomarkers.

DETAILED DESCRIPTION:
Nasal mucus as first line defense barrier of the nasal mucosa contains a variety of proteins that act as functional units. We recently showed that the nasal mucus proteome between allergic rhinitis patients and healthy controls is significantly altered. On protein level, immune response in allergic rhinitis is enhanced and barrier function is reduced as reflected by increased epithelial permeability. Moreover, there is an unfavorable imbalance in innate anti-proteases. Proteases in pollen grain could therefore not be adequately deactivated in the mucus further damaging the epithelium which leads to submucosal penetration of allergens and facilitated presentation to antigen presenting cells.

The aim of the present project is to show changes in nasal mucus proteome between allergic rhinitis patients and healthy controls over the pollen and non pollen season and to further determine whether and if so how the proteome changes under immunotherapy. For the first aim patients and healthy controls will be enrolled at two time points namely during the pollen season and out of the pollen season. Statistical differences will be determined within the groups and between the groups. The protein changes over the time course reflect how allergics but also healthy controls react to allergen challenge. The results should give insight on possible biomarkers that could be used for diagnostics and therapy. Protein substitution or inhibition may be a future therapy to reinforce the barrier function of nasal mucus and treat allergic rhinitis symptoms. The effect of immunotherapy as sole causal therapy will be determined and therapy responders will be compared to non-responders. We hypothesize that responders will show proteome changes similar to healthy conditions. This further concretizes distinct proteins as biomarkers that could be used as therapeutic agents. Moreover proteome changes could be used to predict and monitor therapeutic success or failure and patients may be stratified to be subjected to other therapeutic strategies than immunotherapy saving time and money.

Mucus will be collected with a special suction device equipped with a mucus trap. Then, proteomic analysis will be performed by LC MS/MS mass spectrometry. Database search will identify distinct proteins and their function, origin etc. will be annotated. Protein groups will be analyzed through pathway enrichment and cluster analysis. By this means complex proteomic data can be visualized for a better understanding of global changes in protein networks and functions.

Investigating the nasal mucus proteome in diseased and healthy state leads to a better understanding of its barrier function and reaction to allergens. Distinct proteins and/or proteins groups could be used as biomarkers for novel diagnostic and therapeutic approaches. Furthermore, mechanisms of immunotherapy in responders and success or failure of therapy could be determined.

ELIGIBILITY:
Inclusion Criteria:

* pollen allergy verified by skin-prick test, blood tests for specific IgE (RAST) and allergic rhinitis symptoms, eligible for immunotherapy

Exclusion Criteria:

* chronic infectious diseases, bad overall health condition, pregnancy, long-term intake of nasal and/or systemic steroids or antihistamines, acute and/or chronic rhinosinusitis and parallel participation in other studies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Allergic Rhinoconjunctivitis Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2015-04; Primary Completion 2025-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
AUC of protein spectra obtained by mass spectrometry | 3 years
  Areas under the curve of protein spectra will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- ENT University Hospital Graz, Graz, Styria, Austria

REFERENCES:
- [Background] Tomazic PV, Birner-Gruenberger R, Leitner A, Obrist B, Spoerk S, Lang-Loidolt D. Nasal mucus proteomic changes reflect altered immune responses and epithelial permeability in patients with allergic rhinitis. J Allergy Clin Immunol. 2014 Mar;133(3):741-50. doi: 10.1016/j.jaci.2013.09.040. Epub 2013 Nov 28. PMID 24290289